CLINICAL TRIAL: NCT03115463
Title: Saturation Targets and Resuscitation in Preterm Infants the Delivery Room: A Randomized Controlled Trial
Brief Title: Saturation Targets and Resuscitation in Preterm Trial
Acronym: STARTPreterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Academy of Pediatrics (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Vishal Kapadia, Assistant Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 062014-010; 1K23HD083511-01A1 (NIH)
Record Dates: First submitted 2017-03-14; First posted 2017-04-14 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Oxidative Stress
Keywords: Neonatal Resuscitation; Prematurity; Oxygen
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical care team in the neonatal intensive care unit, investigators running the oxidative stress measurements and investigator assessing neurodevelopmental outcomes will be blinded to which arm the infant was randomized to in the delivery room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OX25 (Experimental): Resuscitation will be initiated at 30% O2. Titration of oxygen during neonatal resuscitation: Intervention is target goal saturations which will be the 10th to 25th percentile saturations observed in healthy term newborns.
  Interventions: Other: Titration of oxygen during neonatal resuscitation
- OX50 (No Intervention): Resuscitation will be initiated with 30% O2 and target goal saturations will be the approximated median SpO2 observed in healthy term newborns as per current NRP guidelines
- OX75 (Active Comparator): Resuscitation will be initiated at 30% O2. Titration of oxygen during neonatal resuscitation: Intervention is target goal saturations which will be the 75th percentile saturations observed in healthy term newborns.
  Interventions: Other: Titration of oxygen during neonatal resuscitation

INTERVENTIONS:
Other: Titration of oxygen during neonatal resuscitation — Resuscitation will be initiated at 30% O2 and target goal saturations will be the 10th to 25th percentile saturations in OX25 and 75th percentile in OX75 group. The control group will be resuscitated with the OX50 strategy in which resuscitation will be initiated with 30% O2 and target goal saturations will be the approximated median SpO2 observed in healthy term newborns as per current NRP guidelines. For the first 6 minutes after birth, target ranges of of all 3 arms are different. After 6 min, the target ranges are are identical.
  Arms: OX25; OX75

SUMMARY:
The purpose of this research project is to determine if use of optimized target oxygen strategy during delivery room resuscitation can reduce oxidative stress in premature newborns. Objective is to compare oxidative stress markers between preterm neonates resuscitated in the delivery room using three different target oxygen strategies. OX50 target oxygen strategy is currently in use and recommended by neonatal resuscitation program. In this strategy oxygen is adjusted to meet the goal transitional saturations which are approximated 50th centile saturations observed in healthy term newborns. In OX25 target oxygen strategy oxygen will be adjusted to meet the goal transitional saturations which are 25th percentile transitional saturations observed in healthy term newborns. In OX75 target oxygen strategy oxygen will be adjusted to meet the goal transitional saturations which are 75th percentile transitional saturations observed in healthy term newborns.

DETAILED DESCRIPTION:
Study Design: A prospective randomized controlled trial of OX50 versus OX25 versus Ox75 will be conducted at Parkland Hospital. This study will test the hypothesis that the OX25 target oxygen strategy will result in successful resuscitation of preterm neonates with less O2 exposure and reduction in oxidative stress compared to the currently recommended Ox50 target O2 strategy and novel OX75 target oxygen strategy.

Study Population: Neonates with obstetric gestational age (GA) of 23-30 weeks, born at Parkland Hospital, Dallas, TX, who require active resuscitation, will be included. Active resuscitation is defined as positive pressure ventilation (PPV), continuous positive airway pressure (CPAP), or ventilation via an endotracheal tube.

Outcomes:

A. Primary outcome:

• Increase in oxidative balance ratio from baseline by 20%.

Sample size and power estimation: The primary outcome for this study is the change from baseline (cord blood - first 2 hour after birth) in the oxidative balance ratio. From our recently completed randomized control trial, mean ∆ oxidative balance ratio for Ox50 in preterm neonates is 9.28 with standard deviation (SD) of 2.42.41 Based on these preliminary data, in order to detect a 20% change in the ∆ oxidative balance ratio, 25 infants are needed for each arm using two sided alpha of 0.05 and power of 80% and allowing 10% attrition.

B. Secondary Outcome:

* Reduction in other oxidative stress markers:
* Reduction in oxygen load in the delivery room
* Time spent in goal saturations
* Time spent with saturations above 94%
* Incidence and frequency of bradycardia during resuscitation
* Incidence of intubation in the delivery room
* Amount of ventilator support needed in the delivery room
* Incidence of neonatal morbidities such as retinopathy of prematurity (ROP), bronchopulmonary dysplasia (BPD), necrotizing enterocolitis (NEC), intraventricular hemorrhage (IVH), periventricular leukomalacia (PVL), neurodevelopmental impairment
* Brain abnormality score on MRI

Study procedure:

A prospective randomized controlled trial of optimal oxygen strategy will be conducted at Parkland Hospital.

Screening procedure: A research nurse will screen and identify eligible mothers admitted to labor and delivery suites at Parkland hospital. Investigators will obtain antenatal informed consent from mothers admitted to the OB service. A total of 75 neonates will be enrolled in the trial, 25 in each group.

Table: Target Oxygen Levels in Blood

Time after Birth OX25 OX50 OX75

1. min 40%-50% 60%-65% 75%-80%
2. min 50%-60% 65%-70% 80%-85%
3. min 60%-70% 70%-75% 85%-90%
4. min 70%-80% 75%-80% 90%-95%
5. min 80%-90% 80%-85% 90%-95%
6. min 85%-95% 85%-95% 90%-95%

10 min 85%-95% 85%-95% 90%-95%

Study intervention and control group: The study intervention #1 is the Ox25 where resuscitation will be initiated at 30% O2 and target goal saturations will be the 25th percentile saturations observed in healthy term newborns.52 The study intervention #2 is the Ox75 where resuscitation will be initiated at 30% O2 and target goal saturations will be the 75th percentile saturations observed in healthy term newborns. The control group will be resuscitated with the OX50 in which resuscitation will be initiated with 30% O2 and target goal saturations will be the approximated median SpO2 observed in healthy term newborns as per current NRP guidelines. Table 1 compare the transitional goal saturations that will be used in OX25, OX50 and Ox75. For the first 6 minutes after birth, target ranges of different strategies are different. After 6 min, the target ranges are similar. Target saturations are an approximation of the percentile curves created by Dawson et al based on transitional saturation data of 306 healthy term neonates who did not receive any intervention other than warmth and stimulation.52

Randomization and Allocation Procedure: Assignment to the OX25, OX50 and OX75 group will use a 1:1:1 allocation ratio. The Biostatistician will use a blocked randomization schema, programmed using SAS Proc Plan (SAS version 9.2, SAS Institute, Cary, NC, USA). Allocation will be concealed by serially numbered, sealed opaque envelopes that will be opened sequentially by the resuscitation team before delivery.

Resuscitation management: The high-risk resuscitation team attends delivery of all neonates < 35 wks GA. Radical pulse oximeters (Masimo, Irvine, CA) will be set to maximal sensitivity with 2 seconds averaging. Randomization will be done before delivery by opening a sealed, opaque envelope. The probe will be placed on the pre-ductal hand within the first 30 seconds of life using previously described strategies to optimize time to reliable signal as per NRP 2011 guidelines. A neonatal transducer (Invos Cerebral Oximeter Monitor , Covidien, Mansfield, Massachusetts) will be attached to left fronto-pareital forehead to measure continuous near infrared spectroscopy (NIRS) measurements. Apart from the randomly assigned O2 strategy, resuscitation will follow 2011 NRP guidelines. Treatment failure will be defined as HR< 60 bpm after 90 seconds of resuscitation. In this event, the O2 concentration will be increased to 100% as recommended by current NRP guidelines. Once HR is stabilized, FiO2 will be reduced to meet the goal saturations of the assigned strategy. If pulse oximetry does not register stable values, resuscitation will be continued at the current FiO2 as long as HR > 100 bpm is maintained. If HR remains below 100 bpm, after making ventilation correcting steps, FiO2 can be increased by 10-20% based on clinician's judgement.

Subsequent NICU management: Following NICU admission, all care decisions including ventilator management will be at the discretion of the attending neonatologist. Target SpO2 will be 88-94% throughout the NICU stay as per unit policy. Infants with O2 requirement at 36 weeks corrected GA will undergo an O2 challenge test to define physiologic BPD as per the NICHD definition.

Collection of baseline variables: Baseline demographic characteristics, maternal and delivery characteristics including maternal age, prenatal clinic attendance, antenatal steroids given, maternal diabetes, illicit drug use, preeclampsia, prolonged rupture of membrane, chorioamnionitis, abruption, previa and cesarean section will be collected. Baseline infant characteristics such as gender, obstetrical GA, birth weight, intrauterine growth restriction, breech presentation, multiple pregnancies, cord blood gas pH, base deficit will be recorded. This data will be collected from the electronic medical records by research nurse and Parkland neonatal intensive care unit database which collects this information on all the infants admitted to Parkland NICU.

Outcomes and Statistical plan by each aim:

A. Specific Aim I: To determine if OX25 will decrease DR O2 load and oxidative stress compared to OX50 and OX75. Investigators hypothesize that OX25 neonates will require less O2 in the DR, spend more time in goal SpO2 range and will have lower oxidative stress

DR O2 exposure and SpO2: SpO2 will be downloaded from pulse oximeters used during resuscitation as per Masimo pulse oximeter guidelines using TRENDCOM software (Masimo, Irvine, CA). Investigators have described and successfully performed acquisition of such data in our previous study. Resuscitation interventions including changes in FiO2 will be recorded at 30 seconds intervals by the OB circulating nurse whose sole responsibility is to record resuscitation details in a pre-specified record sheet as per routine practice at Parkland Hospital.

Oxidative stress and oxidative injury measurement:

Preparation and storage by research nurse: Sample will be centrifuged to separate plasma and stored at -80 C.

A. Oxidative balance ratio: All samples will be analyzed for total hydroperoxides (TH) and biological antioxidant capacity (BAP) using the Free Radical Analytical System (FRAS4 analyzer, H&D SRL, Parma, Italy) as described in our previous study. TH represents the total of radical O2 metabolites produced by peroxidation of protein, lipids and amino acids, measures oxidative damage and serves as a biomarker of overall free radical attack. BAP measures both endogenous and exogenous antioxidative capacity of serum to reduce oxides by inactivating, and eliminating free radicals and reactive O2 species. BAP by exploiting the chemical principle of the well-known ferric reducing ability of plasma provides a reliable measure of biological antioxidant potential of plasma. To estimate the global balance between oxidative stress and antioxidant potential, the oxidative balance ratio (BAP/TH) will be calculated.

B. Other oxidative stress markers: 8-hydroxydeoxyguanosine (8-OHdG), F2-Isoprostanes and Isofurans and Protein Carbonyls. Along with these, investigators will also measure cytokines, Interleukin 1 receptor antagonitst, hyaluronidase.

B. Specific Aim II: Determine if preterm neonates can be resuscitated successfully with less ventilatory support using Ox25. Investigators hypothesize that OX25 infants will achieve quicker heart rate stabilization and will require less ventilatory support including intubation in the DR. Resuscitation interventions including changes in ventilator support, need for CPR will be recorded at 30 seconds intervals by OB circulating nurse whose sole responsibility is to record resuscitation details in a pre-specified record sheet as per the our routine practice. The research nurse will download continuous heart rate data from Masimo pulse oximeters and continuous NIRS data from cerebral oximeter monitor for the duration of resuscitation. Admission parameters will also be recorded by the research nurse.

C. Specific Aim III: Determine if OX25 strategy will result in lower incidence of adverse clinical outcomes compared to OX50 or OX75 strategy. Investigators hypothesize that OX25 neonates will have lower incidence of BPD. Investigators will also record other clinical outcomes such as ROP, NEC, IVH, length of hospitalization, neurodevelopmental impairment and mortality.

Neonatal morbidity during NICU stay: Short term clinical outcomes including duration and type of respiratory support and O2 supplementation during the NICU stay, respiratory morbidities such as respiratory distress syndrome, need for surfactant, pulmonary hypertension, and BPD will be obtained from the NICU database. In addition, other short term morbidities such as sepsis, Grade III/IV IVH, NEC, symptomatic patent ductus arteriosus, severe ROP, length of hospitalization and mortality during NICU stay will also be collected from the NICU database.

Brain MRI at term equivalent age: All study infants who underwent a brain MRI at term equivalent age as part of standard of care at parkland hospital will be assessed for brain abnormality score

Neurodevelopmental impairment: All study infants will follow up at 18-24 months of age in the high risk Low Birth Weight Clinic. A blinded developmental pediatrician will perform standardized neurological examination to identify cerebral palsy. Developmental specialist will administer the Bayley Scale of Infant Development III Instrument. Moderate to severe neurodevelopmental impairment will be defined as Bayley III Motor Developmental Index or Psychomotor Developmental Index score less than 70, moderate or severe cerebral palsy, bilateral blindness, bilateral hearing loss requiring hearing aids or cochlear implants.

ELIGIBILITY:
Inclusion Criteria:

1. Neonates of obstetric gestational age 23-30 weeks
2. Inborn at Parkland Hospital, Dallas, Tx
3. Resuscitation team present to initiate resuscitation

Exclusion Criteria:

1. Prenatally diagnosed cyanotic congenital heart disease
2. Prenatally diagnosed congenital diaphragmatic hernia
3. Prenatally diagnosed significant airway anomaly
4. Prenatally suspected hypoplasia of lungs
5. Preductal saturation cannot be measured
6. Non-viable newborns
7. Prenatally diagnosed condition due to which decision is made to limit resuscitation in the delivery room by parents and neonatologist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Oxidative Balance Ratio from Baseline | within 2 hours after Birth
  Difference in oxidative balance ratio between Cord blood and postnatal sample obtained within 2 hours of life will be assessed.

SECONDARY OUTCOMES:
Reduction in Isoprostane,Isofluran, 8-OHdG and protein carbonyls | Within 2 hours after birth and at 24 hours
  We will measure other oxidative stress markers such as markers of lipid peroxidation: isoprostanes and Isoflurans, measures of oxidative DNA damage: 8-OHdG and Protein carbonyls to assess global oxidative status of the infants
• Reduction in oxygen load in the delivery room | During resuscitation in the delivery room for the first 15 minutes of life
  Oxygen load will be measured for first 15 minutes of life
Time spent in goal saturations | During resuscitation in the delivery room
  Time spent within goal saturation will be presented as percentage of total time
Incidence of bradycardia during resuscitation | During resuscitation in the delivery room
  Bradycardia defined as HR< 100 bpm
intubation in the delivery room | During resuscitation in the delivery room
  Intubation in the delivery room and reason for intubation will be recorded
Grade III/IV Intraventricular hemorrhage | within 6 months
  Defined by Papile classification
Bronchopulmonary dysplasia (BPD) | within 6 months
  Defined by oxygen requirement at corrected 36 weeks gestation
Necrotizing enterocolitis (NEC) | within 6 months
  Defined by modified bell criteria
Retinopathy of prematurity (ROP), necrotizing enterocolitis (NEC), Grade 3/4 intraventricular hemorrhage (IVH), Mortality during NICU stay | Within 1 year
  Defined by operational manual created before the start of the study
Neurodevelopmental Impairment | Within 2 years
  NICHD Neonatal Research Network definition of NDI will be used
Mortality | within 2 years
  Death

CONTACTS AND LOCATIONS:
Overall Officials: Vishal Kapadia, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided